CLINICAL TRIAL: NCT02770963
Title: Efficacy of Acupuncture for Discogenic Sciatica: a Randomized Controlled Trial
Brief Title: Efficacy of Acupuncture for Discogenic Sciatica
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Qin Yao, Postgraduate, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016010401
Record Dates: First submitted 2016-05-05; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Sciatica
Keywords: discogenic; Acupuncture Therapy; randomized controlled trial
MeSH Terms: conditions — Sciatica | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Shenshu (BL23) on bilateral sides and Dachangshu (BL25), Weizhong (BL40), and Chengshan (BL57) on the affected side will be applied.
  Huatuo Brand needle (0.3*75 mm) will be used for BL25 and Huatuo Brand needle (0.3*40mm) will be used for BL23, BL40 and BL57.
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): The acupoints will be the same as the acupuncture group. Specially designed sham needles (0.3*25 mm) will be used . The sham needle consists of a needle handle, needle body, blunt tip and a sterile polyethylene cylindrical foam pad (identical to the pads in the acupuncture group).
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Shenshu (BL23) on bilateral sides and Dachangshu (BL25), Weizhong (BL40), and Chengshan (BL57) on the affected side will be applied.
  A Huatuo Brand needle (0.3*75 mm) for BL25 will be inserted at a depth of 40-70 mm vertically until the patient feels soreness and a distension sensation that radiates to the leg. The needle will be lifted 1-2 mm without rotating or lifting. Huatuo Brand needles (0.3*40 mm) at the other acupoints (BL23, BL40 and BL57) will be inserted 30 mm and manipulated by lifting, thrusting, twirling evenly until the Deqi sensation is achieved. The needles in these acupoints will be manipulated by small evenly applied lifting, thrusting, and twirling movements 3 times every 10 minutes.
  Arms: Acupuncture
Procedure: Sham acupuncture — Specially designed sham needles (0.3*25 mm) will be used. The sham needle consists of a needle handle, needle body, blunt tip and a sterile polyethylene cylindrical foam pad (identical to the pads in the acupuncture group).
  The acupoints will be the same as the acupuncture group. The needle will be inserted vertically until pressed against the skin without penetration. The manipulation will be consistent with the acupuncture group and blind to the patients.
  Arms: Sham acupuncture

SUMMARY:
This trial is designed to evaluate the efficacy of acupuncture on pain relief for patients with discogenic sciatica compared with sham acupuncture.

DETAILED DESCRIPTION:
Background: Sciatica is primarily caused by herniated discs with nerve-root compression. Acupuncture may effectively relieve the pain of discogenic sciatica, but the evidence is limited.

Methods/Design: Sixty patients with discogenic sciatica will be recruited and randomized to receive acupuncture or sham-acupuncture at a 1:1 ratio. Patients in both groups will receive treatment 3 times per week for 4 weeks. The following acupoints will be used: Dachang shu (BL 25), Shenshu (BL 23), Weizhong (BL 40), and Chengshan (BL 57).

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral leg pain diagnosed as discogenic sciatica;
2. Sciatica patients with an average leg pain VAS of 40 mm or higher in the last 24 hours;
3. Aged 18 to 75 years;
4. Leg pains that correlate with CT or MRI findings of lumbar disc herniation;
5. Patients who agree to follow the trial protocol.

Exclusion Criteria:

1. Severe cases with central or giant or ruptured lumbar disc herniation, cauda equina syndrome, foot drop, or surgery requirements;
2. Progressive neurological symptoms after 3 months of strict conservative treatment (e.g., nerve root adhesion, crossed straight-leg testing, or obvious muscle atrophy);
3. Severe cardiovascular, liver, kidney, hematopoietic system diseases, autoimmune diseases, or poor nutritional status;
4. Subjects with cognitive impairment;
5. Pregnancy;
6. Subjects who received acupuncture for sciatica within the past month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
change from baseline in mean weekly VAS of leg pain | Baseline, weeks 1-4, week 16 and week 28
  VAS uses a 100-mm line that is labeled at each end, and 0 mm represents no pain, and 100 mm represents unbearable pain. Patients will rate the VAS (average VAS of leg pain in the past 24 hours), and a researcher will record the VAS once weekly, generally at the third weekly treatment. The mean weekly VAS of leg pain over weeks 1-4 will be calculated as the sum VAS of each week divided by the number of weeks assessed.

SECONDARY OUTCOMES:
Change in mean weekly VAS of low back pain | Baseline, weeks 1-4, week 16 and week 28
  Patients will rate their average low back pain intensity in the past 24 hours using VAS. The mean weekly VAS of low back pain over weeks 1-4 will be calculated as described above for the mean weekly VAS of leg pain over weeks 1-4.
Oswestry disability index | Baseline, week 4, week 16 and week 28
  ODI consists of 10 questions, including pain intensity, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question is scored on a scale of 0-5. The scores for all questions answered are summed and divided by the highest possible score to obtain the index (range 0% to 100%). 0% equals no disability, and 100% is the maximum disability possible
Patients' global impressions of improvement | week 4
  Patients' global impressions of improvement measured using a Likert 7-point scale (higher scores indicate worse outcome).
Patients' expectations for acupuncture | baseline
  This questionnaire includes three brief questions to investigate whether patients believe that acupuncture treatment will help their sciatica. The relationship between patients' expectations and the effectiveness of acupuncture will be investigated because patients' beliefs about treatment enhanced or attenuated the effectiveness of treatment in a previous experimental study .
Blinded evaluation | week 4
  Blinded evaluation as measured by patient questioning of whether they believed they received real acupuncture at week 4. The difference in the proportion of patients who believed that they received real acupuncture between the two groups will be analyzed.
Incidence of serious adverse events | up to 28 weeks
  The investigators will record and evaluate all adverse events .

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yao, Principal Investigator — Department of Acupuncture, Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing (100053), China
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Koes BW, van Tulder MW, Peul WC. Diagnosis and treatment of sciatica. BMJ. 2007 Jun 23;334(7607):1313-7. doi: 10.1136/bmj.39223.428495.BE. No abstract available. PMID 17585160
- [Background] Valat JP, Genevay S, Marty M, Rozenberg S, Koes B. Sciatica. Best Pract Res Clin Rheumatol. 2010 Apr;24(2):241-52. doi: 10.1016/j.berh.2009.11.005. PMID 20227645
- [Background] Ropper AH, Zafonte RD. Sciatica. N Engl J Med. 2015 Mar 26;372(13):1240-8. doi: 10.1056/NEJMra1410151. No abstract available. PMID 25806916
- [Background] Lewis R, Williams N, Matar HE, Din N, Fitzsimmons D, Phillips C, Jones M, Sutton A, Burton K, Nafees S, Hendry M, Rickard I, Chakraverty R, Wilkinson C. The clinical effectiveness and cost-effectiveness of management strategies for sciatica: systematic review and economic model. Health Technol Assess. 2011 Nov;15(39):1-578. doi: 10.3310/hta15390. No abstract available. PMID 22078311
- [Background] Asche CV, Kirkness CS, McAdam-Marx C, Fritz JM. The societal costs of low back pain: data published between 2001 and 2007. J Pain Palliat Care Pharmacother. 2007;21(4):25-33. PMID 18032313
- [Background] Thomas KC, Fisher CG, Boyd M, Bishop P, Wing P, Dvorak MF. Outcome evaluation of surgical and nonsurgical management of lumbar disc protrusion causing radiculopathy. Spine (Phila Pa 1976). 2007 Jun 1;32(13):1414-22. doi: 10.1097/BRS.0b013e318060a5d1. PMID 17545909
- [Background] Ji M, Wang X, Chen M, Shen Y, Zhang X, Yang J. The Efficacy of Acupuncture for the Treatment of Sciatica: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2015;2015:192808. doi: 10.1155/2015/192808. Epub 2015 Sep 6. PMID 26425130
- [Background] Qin Z, Liu X, Wu J, Zhai Y, Liu Z. Effectiveness of Acupuncture for Treating Sciatica: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2015;2015:425108. doi: 10.1155/2015/425108. Epub 2015 Oct 21. PMID 26576192
- [Background] Kreiner DS, Hwang SW, Easa JE, Resnick DK, Baisden JL, Bess S, Cho CH, DePalma MJ, Dougherty P 2nd, Fernand R, Ghiselli G, Hanna AS, Lamer T, Lisi AJ, Mazanec DJ, Meagher RJ, Nucci RC, Patel RD, Sembrano JN, Sharma AK, Summers JT, Taleghani CK, Tontz WL Jr, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of lumbar disc herniation with radiculopathy. Spine J. 2014 Jan;14(1):180-91. doi: 10.1016/j.spinee.2013.08.003. Epub 2013 Nov 14. PMID 24239490
- [Background] MacPherson H, Altman DG, Hammerschlag R, Youping L, Taixiang W, White A, Moher D; STRICTA Revision Group. Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA): extending the CONSORT statement. J Altern Complement Med. 2010 Oct;16(10):ST1-14. doi: 10.1089/acm.2010.1610. PMID 20954957
- [Background] Liu B, Xu H, Ma R, Mo Q, Yan S, Liu Z. Effect of blinding with a new pragmatic placebo needle: a randomized controlled crossover study. Medicine (Baltimore). 2014 Dec;93(27):e200. doi: 10.1097/MD.0000000000000200. PMID 25501074
- [Background] Porchet F, Wietlisbach V, Burnand B, Daeppen K, Villemure JG, Vader JP. Relationship between severity of lumbar disc disease and disability scores in sciatica patients. Neurosurgery. 2002 Jun;50(6):1253-9; discussion 1259-60. doi: 10.1097/00006123-200206000-00014. PMID 12015843
- [Background] Cohen SP, Bogduk N, Dragovich A, Buckenmaier CC 3rd, Griffith S, Kurihara C, Raymond J, Richter PJ, Williams N, Yaksh TL. Randomized, double-blind, placebo-controlled, dose-response, and preclinical safety study of transforaminal epidural etanercept for the treatment of sciatica. Anesthesiology. 2009 May;110(5):1116-26. doi: 10.1097/ALN.0b013e3181a05aa0. PMID 19387178
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Sherman KJ, Cherkin DC, Ichikawa L, Avins AL, Delaney K, Barlow WE, Khalsa PS, Deyo RA. Treatment expectations and preferences as predictors of outcome of acupuncture for chronic back pain. Spine (Phila Pa 1976). 2010 Jul 1;35(15):1471-7. doi: 10.1097/BRS.0b013e3181c2a8d3. PMID 20535051
- [Background] Bartels DJ, van Laarhoven AI, van de Kerkhof PC, Evers AW. Placebo and nocebo effects on itch: effects, mechanisms, and predictors. Eur J Pain. 2016 Jan;20(1):8-13. doi: 10.1002/ejp.750. Epub 2015 Sep 28. PMID 26417885